CLINICAL TRIAL: NCT04562948
Title: Community Applications of the MindShift App
Status: Completed | Type: Observational
Sponsor: University of Windsor (Other)
Collaborators: Anxiety Canada (Unknown)
Responsible Party: Principal Investigator, Lance M. Rappaport, Assistant Professor, University of Windsor
Other Study IDs: MindShift
Record Dates: First submitted 2020-09-11; First posted 2020-09-24 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Anxiety; Depression; Anxiety Generalized; Anxiety Disorders and Symptoms
Keywords: eMental Health; mHealth; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Depression; Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite considerable, replicated evidence of the efficacy and effectiveness of cognitive behavioural therapy, there is an insufficient number of professionals (e.g., psychologists, psychiatrists) in North America to provide evidence-based psychotherapy to all who need it. For example, in light of the COVID-19 pandemic, there is a greater need for resources that are scalable to help a large portion of the public to manage anxiety and attendant psychological distress. One promising avenue to increase the availability of evidence-based mental healthcare relies on technological developments, such as smartphone-enabled apps, to disseminate principles derived from existing evidence-based psychotherapies. However, further research is needed to understand for whom and in what contexts internet- and smartphone-enabled resources are helpful. The present study will examine the utility of one such smartphone enabled app, MindShift, developed by Anxiety Canada in consultation with Canadian and American experts in evidence-based psychotherapy for anxiety disorders. Specifically, the main aim of the present study is to evaluate the effectiveness of the MindShift app to help users manage anxiety and related psychological distress as compared to anxiety and distress prior to app use. Two secondary, exploratory aims of the present study are to examine possible moderators that indicate for whom or in what contexts use of the MindShift app is particularly helpful.

Adult participants 18 years of age and older will be recruited from Canada and the United States of America. Following informed consent, participants will complete baseline assessment of anxiety symptom severity, depressive symptom severity, daily functional impairment, quality of life, alcohol use, use of illicit psychoactive substances, stress associated with the COVID-19 pandemic, and demographic information. Following baseline assessment, participants will be instructed in downloading the MindShift app to their personal mobile phone running either iOS or Android OS software. Participants will then use the MindShift app as they choose for the 16-week duration of the study. Finally, participants will be asked to complete follow-up assessments 2, 4, 8, 12, and 16 weeks following baseline assessment. Follow-up assessments will assess anxiety symptom severity, depressive symptom severity, functional impairment, and quality of life satisfaction on the same measures administered at baseline.

DETAILED DESCRIPTION:
Despite considerable, replicated evidence of the efficacy and effectiveness of cognitive behavioural therapy, there is an insufficient number of professionals (e.g., psychologists, psychiatrists) in North America to provide evidence-based psychotherapy to all who need it. Seminal work from Statistics Canada has emphasized the need for greater access to psychotherapy in Canada. Moreover, in light of the COVID-19 pandemic, there is a greater need for resources that are scalable to help a large portion of the public to manage anxiety and attendant psychological distress. One promising avenue to increase the availability of evidence-based mental healthcare relies on technological developments, such as smartphone-enabled apps, to disseminate principles derived from existing evidence-based psychotherapies. The internet and smartphones provide a novel format to provide information and relevant skills to a large number of users. Recent research indicates that internet-based variants of cognitive behavioural therapy may be efficacious treatments for anxiety and depressive disorders among other conditions. Critically, internet-based treatments are scalable; resources can be provided to many people instantaneously to help them in crises, such as the COVID-19 pandemic. Further study is needed to identify who may benefit from internet-based treatment or require psychotherapy in a more traditional format. For example, whereas mental health professionals receive extensive training in assessment and case formulation to adapt treatments to individuals, internet-based resources are fixed. However, their fixed nature allows internet-based resources to offer a range of tools for users to try in a process of finding those that benefit them in particular situations. Moreover, the ability to access resources on demand presents a unique benefit of internet-based treatments that may support goals of traditional psychotherapy formats to generalize skills into individuals' daily lives. Anxiety disorders are also frequently comorbid with myriad other psychological and psychiatric conditions. Existing treatments for other conditions are often complicated by the presence of a comorbid anxiety disorder, which may be associated with poorer prognosis. Whereas traditional psychotherapy formats consider how to organize treatment for multiple comorbid conditions, internet- and smartphone-enabled resources may help individuals manage concurrent anxiety to support traditional treatment in addressing comorbid conditions. For example, anxiety disorders are often comorbid with substance use disorders; internet- and smartphone-based resources for anxiety disorders may, therefore, supplement existing treatments for substance use disorders for some individuals.

In recent years, there has been a proliferation of smartphone-based apps advertised to help users' mental health and wellness. While many of these apps may use principles of evidence-based treatments, the efficacy, effectiveness, or clinical utility of most apps has not been empirically supported. Overall, internet-based mental health resources may provide useful help to people for whom traditional psychotherapy is not yet available or to augment existing treatment such as through helping to generalize therapeutic skills into one's daily life. However, further research is needed to understand for whom and in what contexts internet- and smartphone-enabled resources are helpful. The present study will examine the utility of one such smartphone enabled app, MindShift, developed by Anxiety Canada in consultation with Canadian and American experts in evidence-based psychotherapy for anxiety disorders. Specifically, the main aim of the present study is to evaluate the effectiveness of the MindShift app to help users manage anxiety and related psychological distress as compared to anxiety and distress prior to app use. Two secondary, exploratory aims of the present study are to examine possible moderators that indicate for whom or in what contexts use of the MindShift app is particularly helpful. Specifically, the research team will examine person-specific and contextual moderators of change over time. For example, the person-specific moderator of baseline anxiety severity may demonstrate a non-linear association with change in anxiety severity over time, which would indicate that the smartphone-based resource is more helpful for individuals in a given range of baseline anxiety severity (e.g., low to moderate) while other treatment formats should be considered for individuals with severe baseline anxiety. Similarly, differences in the rate of anxiety symptom change over time will examine whether use of the app is associated with greater reductions in anxiety and distress when used alone or as an adjunct to traditional psychotherapy or pharmacotherapy. Finally, by examining comorbid conditions and concurrent treatments as moderators of change in anxiety severity over time, the present study will provide some of the first indications of whether use of the MindShift smartphone app to manage anxiety supports existing treatments for conditions frequently comorbid with anxiety disorders.

Adult participants 18 years of age and older will be recruited from Canada and the United States of America using a variety of online platforms and list serves. Following informed consent, participants will complete baseline assessment of anxiety symptom severity, depressive symptom severity, daily functional impairment, quality of life, alcohol use, use of illicit psychoactive substances, stress associated with the COVID-19 pandemic, and demographic information. Following baseline assessment, participants will be instructed in downloading the MindShift app to their personal mobile phone running either iOS or Android OS software. Participants will then use the MindShift app as they choose for the 16-week duration of the study. Finally, participants will be asked to complete follow-up assessments 2, 4, 8, 12, and 16 weeks following baseline assessment. Follow-up assessments will assess anxiety symptom severity, depressive symptom severity, functional impairment, and quality of life satisfaction on the same measures administered at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Canada or the United States of America
* Report any distress related to anxiety
* Are sufficiently comfortable with the English Language to complete study measures
* Have regular access to a smartphone or mobile device that runs the Android or iOS operating systems. This is required to download and use the MindShift app.
* Have semi-regular access to the internet through a computer or mobile device, which is required to complete study assessments.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be adults in Canada and the United States of America recruited through the Anxiety Canada website; advertisements on social media; and email announcements to Canadian and American psychologists and psychiatrists.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Linear and non-linear change in generalized anxiety severity over 16 weeks | 16 weeks
  The Generalized Anxiety Disorder 7-item scale (GAD-7) assesses self-reported severity of generalized anxiety symptoms over the past 2 weeks, specifically symptoms associated with Generalized Anxiety Disorder. The minimum score is 0; the maximum score is 21. Higher scores indicate greater levels of symptom severity. The GAD-7 will be administered at baseline and at 2-, 4-, 8-, 12-, and 16-week planned follow up assessments. The primary outcome measure is linear and non-linear change in generalized anxiety symptom severity over 16 weeks.

SECONDARY OUTCOMES:
Linear and non-linear change in depressive symptom severity over 16 weeks | 16 weeks
  The Patient Health Questionnaire (PHQ-9) assesses self-reported severity of depressive symptoms over the past 2 weeks. The minimum score is 0; the maximum score is 27. Higher scores indicate greater levels of depressive symptom severity. The PHQ-9 will be administered at baseline and at 2-, 4-, 8-, 12-, and 16-week planned follow up assessments. This secondary outcome measure is linear and non-linear change in depressive symptom severity over 16 weeks.
Linear and non-linear change in functional impairment over 16 weeks | 16 weeks
  The Work and Social Adjustment Scale (WSAS) assesses self-reported global functional impairment related to physical and psychiatric distress. The minimum score is 0; the maximum score is 40. Higher scores indicate higher levels of functional impairment related to physical and psychiatric distress. The WSAS will be administered at baseline and at 2-, 4-, 8-, 12-, and 16-week planned follow up assessments. This secondary outcome measure is linear and non-linear change in functional impairment over 16 weeks.
Linear and non-linear change in life satisfaction over 16 weeks | 16 weeks
  The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) assesses one's perceived global quality of life.The minimum score is 16; the maximum score is 80. Higher scores indicate higher levels of life satisfaction. The Q-LES-Q-SF will be administered at baseline and at 2-, 4-, 8-, 12-, and 16-week planned follow up assessments. This secondary outcome measure is linear and non-linear change in life satisfaction over 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lance M Rappaport, Ph.D., Principal Investigator — University of Windsor
Locations (1):
- University of Windsor, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The research team has planned to make data available to other researchers through request to the study principal investigator. Given funding provided by Anxiety Canada and the focused nature of the present study, this IPD plan was considered a careful way to protect potentially identifiable information while limiting the risk that multiple research teams work on identical data analytic projects.

REFERENCES:
- [Background] Andrews G, Basu A, Cuijpers P, Craske MG, McEvoy P, English CL, Newby JM. Computer therapy for the anxiety and depression disorders is effective, acceptable and practical health care: An updated meta-analysis. J Anxiety Disord. 2018 Apr;55:70-78. doi: 10.1016/j.janxdis.2018.01.001. Epub 2018 Feb 1. PMID 29422409
- [Background] Chorpita BF. Modular cognitive-behavioral therapy for childhood anxiety disorders. 2007: Guilford Press.
- [Background] Clark LA, Watson D. Tripartite model of anxiety and depression: psychometric evidence and taxonomic implications. J Abnorm Psychol. 1991 Aug;100(3):316-36. doi: 10.1037//0021-843x.100.3.316. PMID 1918611
- [Background] Forand NR, Huibers MJH, DeRubeis RJ. Prognosis moderates the engagement-outcome relationship in unguided cCBT for depression: A proof of concept for the prognosis moderation hypothesis. J Consult Clin Psychol. 2017 May;85(5):471-483. doi: 10.1037/ccp0000182. Epub 2017 Feb 2. PMID 28150952
- [Background] Grant BF, Stinson FS, Dawson DA, Chou SP, Dufour MC, Compton W, Pickering RP, Kaplan K. Prevalence and co-occurrence of substance use disorders and independent mood and anxiety disorders: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Arch Gen Psychiatry. 2004 Aug;61(8):807-16. doi: 10.1001/archpsyc.61.8.807. PMID 15289279
- [Background] Hasin D, Kilcoyne B. Comorbidity of psychiatric and substance use disorders in the United States: current issues and findings from the NESARC. Curr Opin Psychiatry. 2012 May;25(3):165-71. doi: 10.1097/YCO.0b013e3283523dcc. PMID 22449770
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Kessler RC, Crum RM, Warner LA, Nelson CB, Schulenberg J, Anthony JC. Lifetime co-occurrence of DSM-III-R alcohol abuse and dependence with other psychiatric disorders in the National Comorbidity Survey. Arch Gen Psychiatry. 1997 Apr;54(4):313-21. doi: 10.1001/archpsyc.1997.01830160031005. PMID 9107147
- [Background] Kessler RC, Gruber M, Hettema JM, Hwang I, Sampson N, Yonkers KA. Co-morbid major depression and generalized anxiety disorders in the National Comorbidity Survey follow-up. Psychol Med. 2008 Mar;38(3):365-74. doi: 10.1017/S0033291707002012. Epub 2007 Nov 30. PMID 18047766
- [Background] Khantzian EJ. The self-medication hypothesis of substance use disorders: a reconsideration and recent applications. Harv Rev Psychiatry. 1997 Jan-Feb;4(5):231-44. doi: 10.3109/10673229709030550. PMID 9385000
- [Background] Loucas CE, Fairburn CG, Whittington C, Pennant ME, Stockton S, Kendall T. E-therapy in the treatment and prevention of eating disorders: A systematic review and meta-analysis. Behav Res Ther. 2014 Dec;63:122-31. doi: 10.1016/j.brat.2014.09.011. Epub 2014 Oct 5. PMID 25461787
- [Background] Mohr DC, Burns MN, Schueller SM, Clarke G, Klinkman M. Behavioral intervention technologies: evidence review and recommendations for future research in mental health. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):332-8. doi: 10.1016/j.genhosppsych.2013.03.008. Epub 2013 May 8. PMID 23664503
- [Background] Olthuis JV, Watt MC, Bailey K, Hayden JA, Stewart SH. Therapist-supported Internet cognitive behavioural therapy for anxiety disorders in adults. Cochrane Database Syst Rev. 2016 Mar 12;3(3):CD011565. doi: 10.1002/14651858.CD011565.pub2. PMID 26968204
- [Background] Paschou M, Sakkopoulos E, Tsakalidis A. easyHealthApps: e-Health Apps dynamic generation for smartphones & tablets. J Med Syst. 2013 Jun;37(3):9951. doi: 10.1007/s10916-013-9951-6. Epub 2013 May 12. PMID 23666429
- [Background] Penninx BW, Nolen WA, Lamers F, Zitman FG, Smit JH, Spinhoven P, Cuijpers P, de Jong PJ, van Marwijk HW, van der Meer K, Verhaak P, Laurant MG, de Graaf R, Hoogendijk WJ, van der Wee N, Ormel J, van Dyck R, Beekman AT. Two-year course of depressive and anxiety disorders: results from the Netherlands Study of Depression and Anxiety (NESDA). J Affect Disord. 2011 Sep;133(1-2):76-85. doi: 10.1016/j.jad.2011.03.027. Epub 2011 Apr 14. PMID 21496929
- [Background] Persons JB. Case conceptualization in cognitive-behavior therapy. 1993. In Cognitive therapies in action: Evolving innovative practice. (pp. 33-53). Jossey-Bass.
- [Background] Statistics Canada. Mental health care needs, 2018. 2019; Statistics Canada.